CLINICAL TRIAL: NCT05186740
Title: The ProVee Urethral Expander System Clinical Study
Brief Title: ProVee Urethral Expander System IDE Study (ProVIDE)
Acronym: ProVIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProVerum Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostatic Hyperplasia With Symptomatic Lower Urinary Tract Symptoms
Keywords: BPH / LUTS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized, double-blind, sham-controlled safety and effectiveness study
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject will have noise cancelling headphones on during the treatment. A drape will be placed preventing subjects from observing implant procedure. The follow-up clinic coordinator will not have access to enrolled subjects' medical records including the randomization scheme and treatment procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Device: The ProVee Urethral Expander System (Active Comparator): The ProVee Urethral Expander System consists of two components: a nitinol Expander implant and a 19Fr Delivery System designed to allow the Expander to be deployed under direct vision for the treatment arm.
  Interventions: Device: ProVee Urethral Expander System
- Sham: Ureteroscope and urethral access sheath (Sham Comparator): An ureteroscope housed within the inner lumen of an urethral access sheath will be used under direct vision for the Sham procedure.
  Interventions: Procedure: Urethral Access Sheath
- Crossover ProVee Urethral Expander System (Other): All subjects shall be unblinded following the 3 month follow-up visit. Those subjects randomized to the Sham Arm will be given the opportunity to "crossover" to the ProVee Urethral Expander System.
  Interventions: Device: ProVee Urethral Expander System

INTERVENTIONS:
Device: ProVee Urethral Expander System — ProVee Expander is placed in prostatic urethra to relieve obstruction due to BPH.
  Other Names: ProVee Expander; ProVee
  Arms: Crossover ProVee Urethral Expander System; Device: The ProVee Urethral Expander System
Procedure: Urethral Access Sheath — The Urethral Access Sheath is introduced into the prostatic urethra to simulate the placement of the ProVee Expander.
  Arms: Sham: Ureteroscope and urethral access sheath

SUMMARY:
A study to evaluate the safety, performance, and effectiveness of the ProVee Urethral Expander System (Investigational Device) when used in subjects with symptomatic urinary obstruction related to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, single-blind, sham-controlled study to evaluate the safety, performance, and effectiveness of the ProVee Urethral Expander System (Investigational Device) when used in subjects with symptomatic urinary obstruction related to benign prostatic hyperplasia (BPH). Subjects are assigned to their treatment arm using an unbalanced (2 ProVee:1 Sham) randomization stratified by Investigational Sites.

ELIGIBILITY:
Inclusion Criteria:

1. Males > 45 years of age
2. IPSS of ≥ 13, IPSS V/S > 1 at baseline assessment
3. Prostate volume of ≥ 30 cc and ≤ 80 cc
4. Prostatic urethral L2 lengths ≥ 3.75cm by TRUS
5. Failed, intolerant, or subject choice to not take a medication regimen for the treatment of LUTS

Exclusion Criteria:

1. Void volume <125 ml; Qmax > 12ml/s; PVR > 250 ml
2. Obstructive median lobe defined by EITHER (>10mm protrusion on sagittal mid-prostate plane as measured by TRUS) OR an obstructive median lobe seen on cystoscopy e.g., 'ball valve''
3. High bladder neck, with the absence of lateral lobe encroachment indicating a high likelihood of primary bladder neck obstruction
4. Anatomy that would prevent the apices of the ProVee from engaging with the lateral lobes e.g., high degree of bladder neck angulation such that the anterior bladder neck is not visible
5. Acute urinary retention
6. Known immunosuppression
7. History of or suspected prostate or bladder cancer
8. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer (Subjects with a PSA level above 2.5 ng/mL, or age specific, or local reference ranges should have prostate cancer excluded to the Investigator's satisfaction, including a SOC biopsy if indicated).
9. Recent urinary tract stones, OR widespread calcifications on the prostatic urethral wall, within 3 months of index procedure
10. A history of prostatitis within the last two years
11. Active or history of epididymitis within the past 3 months
12. Neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes'
13. History of urinary retention within 12 months of baseline assessment
14. Requiring self-catheterization to void
15. An active urinary tract infection (UTI) at time of index procedure
16. Gross haematuria, within 3 months of index procedure
17. Subjects with known allergy to nickel or titanium
18. Life expectancy estimated to be less than 60 months
19. Taking androgens, unless eugonadal state for at least 3 months or greater with a stable dosage for at least 2 months as documented by the Investigator
20. Use of 5-alpha-reductase inhibitors (e.g., dutasteride, finasteride) within 6 months of baseline assessment
21. Use of Phenylephrine / Pseudoephedrine within 24 hours of baseline assessment
22. Use of alpha-blockers (e.g., Terazosin, Doxazosin, Alfuzosin, Tamsulosin) within 2 weeks of baseline assessment
23. Use of estrogen or drug-producing androgen suppression (e.g. gonadotropin-releasing hormonal analogues) within 1 year of baseline assessment
24. Use of antihistamines, anticonvulsants, and antispasmodics within 1 week of baseline assessment unless there is documented evidence that the patient was on the same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study)
25. Use of anticholinergics or cholinergic medication within 2 weeks of baseline assessment
26. Use of beta-blockers where the dose is not stable. (Stable dose is defined as having the same medication and dose in the last 6 months)
27. Use of Phosphodiesterase-5 Enzyme Inhibitors in doses for BPH within 2 weeks of baseline assessment
28. Current treatment with anticoagulants (e.g., warfarin or enoxaparin) or antiplatelet medications other than aspirin (e.g., clopidogrel, or alternative and ASA). Patient unable to stop taking antiplatelet and/or antiplatelets within 3 days prior to the procedure or warfarin at least 5 days prior to the procedure. Low dose aspirin ≤100mg/day not prohibited
29. Future fertility concerns
30. Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate; including penile implants
31. Previous pelvic irradiation or radical pelvic surgery
32. Previous rectal surgery (other than hemorrhoidectomy) or known history of rectal disease
33. Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
34. Urethral pathologies that may prevent insertion of Delivery System
35. Uncontrolled diabetes mellitus including Hgb AIC >8%
36. Overactive bladder (OAB) requiring treatment by OAB medication
37. Urinary incontinence
38. Patients taking tri-cyclic antidepressants.
39. Compromised renal function (i.e., serum creatinine >1.8 mg/dl or upper tract disease)
40. Hepatic disorder, bleeding disorders or metabolic impairment that might confound the results of the study or have a risk to subject per investigator's opinion
41. Any major comorbidities or presence of unstable conditions, e.g., uncontrolled HTN, NYHA Class III or IV, cardiac arrhythmias that are not controlled by medication/medical device, myocardial infarction within the past 6 months, COPD with FEV1 <50, renal illness that might prevent study completion or would confound study results
42. Vulnerable populations such as incarcerated or institutionalized adults, inmates, patients with physical, psychological (such as developmentally delayed adults), or medical impairment that might, in the judgment of the Investigator, prevent study completion or comprehension, or may confound study results (including patient questionnaires)
43. History or current medical condition that would result in an unacceptable patient risk if that subject were to be included in the study
44. Any subject that is currently enrolled in another ongoing investigational study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 221 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Golden State Urology, Sacramento, California
  - Urological Research Network Corp, Hialeah, Florida
  - Advanced Urology Institute, Palm Coast, Florida
  - Tampa Urology LLC, Tampa, Florida
  - Avant Concierge Urology, Winter Garden, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Sheldon Freedman MD, Las Vegas, Nevada
  - Mount Sinai, New York, New York
  - Manhattan Medical Research Practice, New York, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Midtown Urology Assoc., Austin, Texas
  - Urology Austin, Austin, Texas
  - Houston Methodist, Houston, Texas
  - Urology of Virginia, Virginia Beach, Virginia
- University Health Network, Toronto, Ontario, Canada
- St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ProVerum Website — https://www.proverummedical.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All primary endpoint results are now entered. This Clinical Study Protocol and Statistical Analysis Plan has been redacted in accordance with the regulations at 42 CFR 11.48(a)(5). All SAEs reported have been adjudicated by CEC as not device or procedural related.
Period: Overall Study
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath
Started | 150 | 71
Sham Participants Crossed Over to Device at 3 Month Follow-up | 0 | 64
Completed | 150 (ITT Analysed) | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: At the 3 month follow up, there were 64 participants crossed over from Sham (Ureteroscope and Urethral Access Sheath) Arm/Group to receive the device (ProVee Urethral Expander System)
Groups:
- Total: Total of all reporting groups
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Total
Number analyzed (Participants) | 150 | 71 | 221
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 64.0 (8.7) | 64.5 (8.2) | 64.2 (8.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 150 | 71 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 6 | 25
  Not Hispanic or Latino | 128 | 63 | 191
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Device or Procedure Related Serious Adverse Events (Time Frame: Procedure to 12 Months)
Description: This includes the rate of device or procedure related serious adverse events
Time Frame: Procedure - 12 months
Population: At 3 month follow-up visit, 64 subjects were crossed over from Sham (Uretheroscope and urethral access sheath) to Device (The ProVee Urethral Expander System)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Crossover ProVee Urethral Expander System
Number analyzed (Participants) | 150 | 71 | 64
Participants | 0 | 0 | 0

2. Primary Outcome: Safety: Number of Participants With Need for Urinary Catheterization (Time Frame: >7 Days Post Procedure)
Description: The rate of extended post-operative urinary catheterization for inability to void among patients treated with the ProVee device.
Time Frame: 7 days post treatment through to 12 months
Population: At 3-month follow up, 64 subject were crossed over from Sham (Ureteroscope and Urethral Access Sheath) to Device (The ProVee Urethral Expander System).
Measure: Count of Participants; unit: Participants
Groups:
- Device: The ProVee Urethral Expander System: he ProVee Urethral Expander System consists of two components: a nitinol Expander implant and a 19Fr Delivery System designed to allow the Expander to be deployed under direct vision for the treatment arm.
  ProVee Urethral Expander System: ProVee Expander is placed in prostatic urethra to relieve obstruction due to BPH
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Crossover ProVee Urethral Expander System
Number analyzed (Participants) | 150 | 71 | 64
Participants | 0 | 0 | 0

3. Primary Outcome: Effectiveness: Number of Participants With Reduction in BPH Symptoms Compared to Sham (Time Frame: Procedure to 3 Months)
Description: The ProVee Treatment Group will be considered superior to the Sham Treatment Group when the mean 3-month improvement from baseline score for the IPSS symptom questionnaire demonstrates a minimum statistical margin of 25% compared to mean improvement from baseline for the Sham Treatment Group alone.
Time Frame: Procedure to 3 months
Population: Following the 3 month follow up, 64 subjects were crossed over from sham (ureteroscope and urethral access sheath) to device (the ProVee ureteral expander system)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Crossover ProVee Urethral Expander System
Number analyzed (Participants) | 150 | 71 | 64
Participants | 0 | 0 | 0

4. Primary Outcome: Effectiveness: Number of Participants With Symptoms Improvements (Time Frame: Procedure to 12 Months)
Description: The mean percent change in IPSS in the treatment arm is at least 30% improvement over the patient's pre-treatment baseline score.
Time Frame: Procedure to 12 months
Population: Following the 3 month follow up, 64 subjects from sham (ureteroscope and urethral access sheath) crossed over to device (the ProVee urethral expander system)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Crossover ProVee Urethral Expander System
Number analyzed (Participants) | 150 | 71 | 64
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All subjects are followed for 3 months until the co-primary effectiveness endpoints are evaluated. After their 3-month visit, all subjects are unblinded to their treatment assignment. Subjects assigned to the ProVee Device will continue to be followed up to 60 months post implantation. Following unblinding, subjects assigned to the control arm may (crossover to the active treatment). After being treated, Crossover Subjects will be followed using the same schedule used with the ProVee Device.
Description: Same
Arm/Group | Device: The ProVee Urethral Expander System | Sham: Ureteroscope and Urethral Access Sheath | Crossover ProVee Urethral Expander System
All-Cause Mortality (participants affected / at risk) | 1/150 | 0/71 | 0/64
Serious Adverse Events (participants affected / at risk) | 8/150 | 0/71 | 0/64
Other Adverse Events (participants affected / at risk) | 1/150 | 0/71 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: The ProVee Urethral Expander System (N=150) | Sham: Ureteroscope and Urethral Access Sheath (N=71) | Crossover ProVee Urethral Expander System (N=64)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Small bowel obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Cerebrovascular accident (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — This serious adverse event has not been adjudicated by CEC as device or procedural related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: The ProVee Urethral Expander System (N=150) | Sham: Ureteroscope and Urethral Access Sheath (N=71) | Crossover ProVee Urethral Expander System (N=64)
Dry Mouth (General disorders) | 1 (1) | 0 (0) | 0 (0) — This adverse event was adjudicated by the CEC as not device or not procedural related.

LIMITATIONS AND CAVEATS:
This Clinical Study Protocol and Statistical Analysis Plan has been redacted in accordance with the regulations at 42 CFR 11.48(a)(5). Note that the all cause mortality results, the CEC adjudicated that the death was related to a pre-existing condition. For the serious adverse events, no reported serious adverse events have been adjudicated by CEC as device or procedural related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT05186740/Prot_SAP_005.pdf